CLINICAL TRIAL: NCT00471783
Title: The Effects of Flossing With a Chlorhexidine Solution on Interproximal Gingivitis: a Randomized Controlled Trial
Brief Title: Flossing With Chlorhexidine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Foundation for Dental Hygiene Research and Education (Other); British Columbia Dental Hygienists' Association (BCDHA) (Industry)
Responsible Party: Dr. Donald Brunette, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H05-70513
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Gingivitis
Keywords: gingivitis; chlorhexidine; dental floss; RCT; bleeding on probing; gingival and plaque indices
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Chlorhexidine is the generic name of the mouthwash, Peridex is the brand name.

SUMMARY:
To determine if flossing with a dental floss presoaked in chlorhexidine, an anti-microbial mouth wash, would improve the clinical signs of gingivitis, an inflammation of the gums characterized by red, swollen, bleeding gums. And to determine if applying chlorhexidine via dental floss would result in tooth staining, which is common with chlorhexidine mouthwashes.

DETAILED DESCRIPTION:
Purpose of study: To determine if dental floss presoaked in 0.12% chlorhexidine is more effective at reducing the signs of gingivitis, such as bleeding, than a dental floss in placebo solution of 0.1% quinine sulphate.

Trial design: The study will consist of a double-blinded, placebo-controlled parallel three-month clinical trial.

Randomization of subjects into study groups: Subjects randomized with a computer-generated randomization table and balanced block design to make the two groups equal in number of subjects.

Trial schedule:

1. Screening for potential subjects & consent obtained. Calibration of examiner.
2. Week -1: Professional prophylaxis consisting of scaling and polishing.
3. Week 0: Baseline data (GI, SI, PI, BOP, PD) collected on subjects enrolled into the study. OHI - flossing. Subject randomized into a study group.
4. Week 6: Subjects reassessed for GI, SI, PI, BOP, PD. Compliance check. Replenish floss supply. Subject concerns or questions addressed.
5. Week 12: Subjects reassessed for GI, SI, PI, BOP, PD. All floss boxes and logbook returned. Subject concerns or questions addressed. Subject exited from study and returned to the care of his or her regular dental professional.

Measurements for data collection (done in this order):

1. Gingival index (GI) (modification of Löe & Silness, 1963)
2. Stain Index (SI)
3. Plaque index (PI) (modification of Silness and Löe, 1964)
4. Bleeding on Probing (BOP)
5. Probing Depth (PD)

ELIGIBILITY:
Inclusion Criteria:

To be considered for inclusion into the study, subjects must fulfill the following conditions:

* 18 years and older
* Have gingivitis (i.e., have pocket depths of 4 mm or less), but not periodontitis
* Willing to floss every day and have the necessary dexterity to floss
* Have a minimum of 20 natural teeth, including 4 molars
* Have at least 10 bleeding sites
* Be a non-smoker

Exclusion Criteria:

Subjects will be excluded from the study, if they have any of the following conditions:

* Pregnant or plan to be pregnant within the next 3 months
* Allergic to chlorhexidine or quinine sulphate
* Require pre-medication with antibiotics for dental treatment
* Currently taking antibiotics
* Currently taking Dilantin, Cyclosporin A, Nifedipine or other calcium channel blockers, aspirin or anti-coagulants
* Currently using chlorhexidine or whitening products
* Have active carious lesions
* Have orthodontic braces
* Have more than 2 crowns or bridges
* Have more than 2 implants
* Have full or partial dentures
* Have periodontitis, i.e., pocket depths of 5 mm or more in more than 2 sites in the mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine if dental floss presoaked in 0.12% chlorhexidine is more effective at reducing the signs of gingivitis, such as bleeding, than a dental floss in placebo solution of 0.1% quinine sulphate. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Brunette, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Dr. Ian Low, 2031 West 41st Avenue, Vancouver, British Columbia, Canada